CLINICAL TRIAL: NCT01669707
Title: Endostar Durative Transfusion Combining With Gemcitabine-Cisplatin to Treat Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Liyan Xu, Chief of Medical Oncology Department, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingCH001
Record Dates: First submitted 2012-08-13; First posted 2012-08-21 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Endostar; advanced Non-small cell lung cancer; Continued Pumping into vein; Gemcitabine; Carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endostar -Continued Pumping into+GP (Experimental): Endostar that is Continued Pumping into vein Combining With Gemcitabine -Cisplatin
  Interventions: Drug: Endostar -Continued Pumping into+GP
- Endostar -injecting into +GP (Active Comparator): Endostar that is injecting into vein with Gemcitabine -Cisplatin
  Interventions: Drug: Endostar -injecting into +GP

INTERVENTIONS:
Drug: Endostar -Continued Pumping into+GP — Gemcitabine(G):1000mg/m2 intravenous injection on d1,8 q3w; Cisplatin (P):75mg d1 q3w; Endostar:7.5 mg/m2 Continued Pumping into vein with saline,Each pump use 120 hours and the dosage is 7.5mg/m2*5 ,on day 1 to day 14, discontinuancing for 7 days and 21 days is one cycle,Continued using 2-4cycles.
  Arms: Endostar -Continued Pumping into+GP
Drug: Endostar -injecting into +GP — Gemcitabine(G):1000mg/m2 intravenous injection on d1,8 q3w; Cisplatin (P):75mg iv on d1 q3w; Endostar:7.5 mg/m2 injecting into vein for 4 hours with saline on day 1 to day 14, discontinuancing for 7 days and 21 days is one cycle.Continued using 2-4cycles
  Arms: Endostar -injecting into +GP

SUMMARY:
The purpose of this study is to determine whether Endostar pumping into vein with Gemcitabine-Cisplatin are more effective than Endostar with Gemcitabine-Cisplatin regularly in the treatment of Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Endostar have anti-tumor activity by against vascular endothelial growth factor for initial treatment. This study was designed to evaluate the safety and efficacy of Endostar Continued vein-pumping Combining with Gemcitabine-Cisplatin (GP)chemotherapy in patients with NSCLC,and seeking for more effective injection.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed NSCLC;
2. primary treatment,inoperable stage IIIB/IV NSCLC;
3. Age of 18-75years; Gender Not Required;
4. Adequate hematologic, renal, and hepatic function ,Specific index as follows:

   liver function: S-Bilirubin ≤1.5 ULN ; Transaminase≤2 ULN. renal function: S-Creatinine ≤1.2 ULN; blood urea nitrogen ≤1.2 ULN . ULN: upper normal limit. Marrow Hemopoietic Function: WBC≥4.0×10^9/l, ANC≥2.0×10^9/l platelet count ≥100×10^9/l, Hb≥100 g/l;
5. ECOG PS 0-2,Life expectancy ≥ 3 months; endure more than two cycle chemotherapy;
6. The patients have explicit lung tumor lesions and the lesions were measurable; (According to the standard of RECIST1.1, they should have at least one of accurately measurable lesions with the largest diameter ≥ 10mm by spiral CT, MRI);
7. No history of serious drug allergy;
8. Informed consent should be obtained before treatment.

Exclusion Criteria:

1. Symptomatic brain metastases with cognitive disorder,bone metastases with complications;
2. Major organ dysfunction and Serious Heart Disease( congestive heart-failure,incontrollable high-risk arrhythmia,unstable angina, valvular disease, myocardial infarct and Resistant hypertension,);
3. Serious complications and investigator consider it is unsuited enrolling;
4. Pregnant or lactating women;
5. Allergic to research drug;
6. participating in other experimental trials and receive the treatment in four weeks;
7. The position that is for observing curative effect have a radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-04 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | two years

SECONDARY OUTCOMES:
Overall survival (OS) | two years
Clinical benefit rate (CBR) | two years
Number of Participants With Adverse Events(AE) as a Measure of Safety and Tolerability | two years

CONTACTS AND LOCATIONS:
Locations (1):
- The Beijing Chest Hospital, Beijing, China